CLINICAL TRIAL: NCT02519998
Title: Tissue Repository and Master Database for Concussion Biomarker and Risk Calculator Development
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Collaborators: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: 14D.611
Record Dates: First submitted 2015-03-25; First posted 2015-08-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Brain Concussion
Keywords: Biomarkers; Electrocardiography; Balance; Neuropsychiatric assessment; Cortisol; Calcitonin-gene-related peptide; Electroencephalography; Optical coherence tomography; Von Frey Testing
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine Blood Saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Concussed patients: The clinical focus of this study will be on concussed athletes, both children and adults, and we will also include non-sports patients who have mild traumatic brain injury due to other situations including slip and fall, occupational, motor vehicle accidents, assault, and blast exposure.
  Interventions: Other: Concussion
- Non-concussed patients: Cohort control. Primarily athletes who undergo routine pre-season baseline assessment

INTERVENTIONS:
Other: Concussion — Study groups are differentiated based on presence of concussion. No intervention is being made in either population (observational study)
  Groups: Concussed patients

SUMMARY:
The purpose of this study is to prospectively collect a comprehensive, multi-modality set of diagnostics on patients who have had a concussion, repeating some of these tests serially over time, so that the investigators may then in the future perform retrospective data mining to determine if there were a biomarker or risk calculator that could be used to guide return-to-play and other medical decisions.

DETAILED DESCRIPTION:
Concussions comprise a type of mild traumatic brain injury in which mechanical forces disrupt brain metabolism causing transient neurological symptoms.

At the current time, there is no universally agreed-upon objective biomarker or risk calculator of concussion upon which physicians can prognosticate future risk, identify optimal treatments, and for sports medicine physicians, decide if and when a particular player were safe to be returned to play.

While the majority of patients experience a full recovery within a few weeks of a concussion, several going on to have chronic, debilitating symptoms, and all patients experience a permanently increased risk of experiencing more debilitating and long-lasting symptoms with each subsequent concussion. For certain people with certain genetic (e.g., ApoE status) and psychosocial (e.g., alcohol abuse, depression) risk factors, even a single concussion can put them at greater risk for earlier and more severe forms of dementia decades hence.

The purpose of this study is to prospectively collect a comprehensive, multi-modality set of diagnostics on patients who have had a concussion, repeating some of these tests serially over time, so that the investigators may then in the future perform retrospective data mining to determine if there were a biomarker or risk calculator that could be used to guide return-to-play and other medical decisions.

This study plans to collect biological specimens (blood, saliva, urine, hair follicles), electrophysiological (EEG, EKG), imaging (HCT, MRI, PET, SPECT), ambulatory (actigraphy), sensory thresholds (Von Frey), ophthalmologic (fundoscopic photographs, OCT, SSVEPs), vestibular (ENG, BESS, BioSway) along with demographic, medical history, medication, psychosocial data and the results on validated instruments of cognition, mood, sleep, head discomfort and quality of life.

Because it is important to determine the variability not only within the concussion group but also between groups, the investigators will also recruit a control cohort, specifically athletes who are already undergoing baseline cognitive testing pre-season. The clinical focus of this study will be on concussed athletes, both children and adults, and the investigators will also include non-sports patients who have mild traumatic brain injury due to other situations including slip and fall, occupational, motor vehicle accidents, assault, and blast exposure.

ELIGIBILITY:
Inclusion Criteria:

* All patients, 10 years of age or older with concussion being evaluated at the Jefferson Comprehensive Concussion Center in Philadelphia, PA, or by Jefferson Comprehensive Concussion Center physicians at other locations (including Rothman Institute sports medicine clinics in Bryn Mawr, PA, Marlton, NJ, Washington Township, NJ). The target population will be those with suspected concussions.

Exclusion Criteria:

* Patients not presenting at the Jefferson Comprehensive Concussion Center or affiliated locations.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals ages 10 or older. If the patient has experienced a suspected concussion, must be a patient at the Jefferson Comprehensive Concussion Center.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Medical history indicative of concussion | Upon enrollment
  Basic medical history demographics gathered during patient's regular clincal visit.

SECONDARY OUTCOMES:
Neurocognitive Testing and Assessment Batteries | 1 year
  Sports Concussion Assessment Tool (SCAT-3)
Neurocognitive Testing and Assessment Batteries | 1 year
  Balance Error Scoring System (BESS)
Neurocognitive Testing and Assessment Batteries | 1 year
  King Devick Test
Neurocognitive Testing and Assessment Batteries | 1 year
  Acute Concussion Evaluation (ACE)
Neurocognitive Testing and Assessment Batteries | 1 year
  Beck Depression Inventory (BDI)
Neurocognitive Testing and Assessment Batteries | 1 year
  Beck Anxiety Inventory (BAI)
Neurocognitive Testing and Assessment Batteries | 1 year
  World Health Organization-Five Well-being Index (WHO-5)
Neurocognitive Testing and Assessment Batteries | 1 year
  Multidimensional Anxiety Scale for Children (MASC)
Neurocognitive Testing and Assessment Batteries | 1 year
  Spence Children's Anxiety Scale
Neurocognitive Testing and Assessment Batteries | 1 year
  "SCARED" Montgomery-Åsberg Depression Rating Scale
Neurocognitive Testing and Assessment Batteries | 1 year
  ImPACT
Neurocognitive Testing and Assessment Batteries | 1 year
  Trails A and B Forward
Neurocognitive Testing and Assessment Batteries | 1 year
  Reverse Digit Span
Neurocognitive Testing and Assessment Batteries | 1 year
  Jefferson After Concussion Test (JACT)
Neurocognitive Testing and Assessment Batteries | 1 year
  Rivermead Post Concussion Symptom Questionnaire (RPQ)
Neurocognitive Testing and Assessment Batteries | 1 year
  Traumatic Brain Injury-Quality of Life (TBI-QOL)
Neurocognitive Testing and Assessment Batteries | 1 year
  Mayo-Portland Adaptability Inventory (MPAI-4)
Neurocognitive Testing and Assessment Batteries | 1 year
  Migraine Disability Assessment (MIDAS)
Neurocognitive Testing and Assessment Batteries | 1 year
  Fatigue Severity Scale
Neurocognitive Testing and Assessment Batteries | 1 year
  Epworth Sleepiness Scale
Neurocognitive Testing and Assessment Batteries | 1 year
  Pittsburgh Sleep Quality Index
Diagnostic Procedures | 1 year
  Galvanic skin response
Diagnostic Procedures | 1 year
  Electrocardiography (EKG)
Diagnostic Procedures | 1 year
  Electroencephalography (EEG)
Diagnostic Procedures | 1 year
  Fundoscopy Optical Coherence Tomography (OCT)
Diagnostic Procedures | 1 year
  Von Frey Sensory Filament Thresholds
Diagnostic Procedures | 1 year
  BioSway
Biospecimens | 1 year
  Blood
Biospecimens | 1 year
  Siliva
Biospecimens | 1 year
  Urine
Clinically Acquired Imaging | 1 year
  CT, MRI
Opthalmologic | 1 year
  Fundoscopic photographs
Opthalmologic | 1 year
  Optical coherence tomography
Tactile Sensation | 1 year
  Von Frey sensory thresholds

CONTACTS AND LOCATIONS:
Overall Officials: Mijail Serruya, MD, PhD, Principal Investigator — TJUH
Locations (1):
- Jefferson Comprehensive Concussion Center, Philadelphia, Pennsylvania, United States